CLINICAL TRIAL: NCT05563675
Title: Comparing Morning and Evening Dosing of Inhaled Long-Acting Muscarinic Antagonists for the Prevention of Hospitalization Requiring AECOPD or Death from All Causes - the LAMA by Night Study Utilizing a Comprehensive Nationwide Digital Platform for Recruitment Into a Pragmatic Randomized Controlled Trial Integrated with National Registries to Follow Outcomes
Brief Title: Once Daily Long-Acting Muscarinic Antagonists Administered in the Evening for Prevention of Chronic Obstructive Pulmonary Disease Exacerbations Requiring Hospitalization or Death from Any Cause
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol_LAMA
Record Dates: First submitted 2022-09-23; First posted 2022-10-03 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: COPD Exacerbation
Keywords: LAMA; Bedtime administration

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to one of two treatment strategies by computer-generated allocation, to either LAMA administration in the morning or evening. Randomization groups will be allocated according to a computer-generated randomization. Data will be entered by participants directly into REDCap questionnaires. Consent and randomization will take place on day 0. The result of the randomization will be shown directly to the participant on their screen and sent to the participant's official electronic mailbox.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators will be blinded for the treatment allocation, but the trial participants will not be blinded. However, since all endpoints are assessed using prespecified registry-based definitions, bias should be negligible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning administration of LAMA (No Intervention): Participants randomized to this group (with or without the combination of ICS and/or LABA) will be instructed to take their LAMA as usual in the morning between 6 and 12am.
- Bedtime administration of LAMA (Experimental): Participants randomized to this group (with or without the combination of inhaled corticosteroids (ICS) and/or long-acting beta2-agonists (LABA)) will be instructed to take their LAMA-containing inhalation between 8pm. and 2am.
  Interventions: Drug: Long acting muscarinic antagonists (LAMAs) in the evening

INTERVENTIONS:
Drug: Long acting muscarinic antagonists (LAMAs) in the evening — LAMAs administered at bedtime (8pm - 2am)
  Arms: Bedtime administration of LAMA

SUMMARY:
To examine, among once-daily LAMA using COPD patients, whether evening administration of LAMA is superior with respect to the incidence of hospitalization requiring AECOPD or death from all causes than the more conventional morning administration.

DETAILED DESCRIPTION:
One of the most feared complications associated with chronic obstructive pulmonary disease (COPD) is acute exacerbation (AECOPD). On average, each COPD patient experiences 0.5 to 3.5 acute exacerbations per year, which is an important reason for the hospitalization, disease progression and mortality as well as decline in health status and lung function(1,2).

Treatment with a long-acting muscarinic antagonist (LAMA) reduces dyspnoea and the risk of exacerbations in patients with COPD by binding to muscarinic receptors in bronchial smooth musculature and thus inhibiting cholinergic bronchial constriction. LAMAs are given as inhalation therapy once daily (most often) or twice daily(3).

Most COPD-patients experience their worst symptoms and experience exacerbations in early morning hours, before getting out of bed(4). This might be explained by the physiological diurnal changes in the activity of the parasympathetic homeostasis system since this is most active at night to improve digestion and other secretions(5).

Correspondingly, the activity of the sympathetic system is physiologically suppressed at night, and stimulation of β-2 receptors is thus also low (and opposite for M-3 receptors). Taken together, the balance of sympathetic-parasympathetic tone is shifted significantly towards the latter. Most available LAMA treatments are dosed once daily in the morning.

Thus, for a COPD patient, being at a trough level of LAMA (which antagonizes the para-sympathetic system) at late night/early morning, may carry a hazard for the patient.

Studies have found that lung function measured as forced expiratory volume in 1 second (FEV1) improvement peaks approximately 2 hours after LAMA administration, and that FEV1 is still significantly improved at 7 hours post treatment but decreases towards the trough level of the LAMA(6). However, as a corollary to the above, when the medicine is probably most needed (02.00 a.m. to 07.00 a.m.), the effect is at its lowest level, which may not be desirable, since a low effect of the most important preventive medicine against AECOPD at this time, may lead to more exacerbations.

Evening administration, on the contrary, would lead to a greater and more certain effect regarding bronchodilation and reduced secretion in the early morning hours, and a maximum effect should be expected during the entire night.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than or equal to 30 years
2. Current treatment with LAMA once daily (as recorded in the Danish National Prescription Registry and confirmed by the participant via questionnaire)
3. Self-reported COPD

Exclusion Criteria:

1. Patients who decline to participate.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10011 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
COPD-related hospitalization-requiring (severe) exacerbations | 12 months from randomization
All-cause mortality | 12 months from randomization

SECONDARY OUTCOMES:
Moderate, non-hospitalization-requiring COPD exacerbations | 12 months from randomization
Number of admissions for all causes | 12 months from randomization
Number of admissions in the intensive care unit (ICU) for all causes | 12 months from randomization
Number of admissions requiring non-invasive ventilation (NIV) treatment | 12 months from randomization
Mortality (all-cause) | 12 months from randomization
Use of short-acting β2-agonists (SABA); pick-up rate | 12 months from randomization
  Data collected from the Danish National Prescription Registry
Change in COPD assesment test (CAT) score | 12 months from randomization
  Measured by questionnaire at 6 and 12 months post-randomization. Measured on a scale from 0 to 40. Score of 0-9 means low impact of COPD and score of 31-40 means very high impact.
Change in medical research council (MRC) score | 12 months from randomization
  Measured by questionnaire at 6 and 12 months post-randomization. Measures baseline functional disability due to dyspnoea on a scale from 0 to 5, 0 meaning no disability and 5 meaning significant disability due to COPD.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev-Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Both negative, positive, and inconclusive results will be submitted for publication in peer-reviewed journals and presented at international scientific conferences.
  Participant-level data and statistical code will not be published.

REFERENCES:
- [Derived] Sivapalan P, Romer V, Jordan A, Johansen ND, Pareek M, Modin D, Mathioudakis AG, Vestbo J, Vognsen AK, Eklof J, Hurst JR, Klausen TW, Biering-Sorensen T, Jensen JS. Evening administration of long-acting muscarinic antagonists in COPD - a randomized controlled trial. BMC Pulm Med. 2025 Dec 3;25(1):552. doi: 10.1186/s12890-025-03952-y. PMID 41340061
- [Derived] Sivapalan P, Romer V, Wirenfeldt Klausen T, Dyrby Johansen N, Pareek M, Modin D, Mathioudakis A, Vestbo J, Eklof J, Jordan A, Hurst JR, Biering-Sorensen T, Jensen JU. AM/PM dosing of LAMA for COPD: a randomized controlled trial protocol using digital recruitment and registries. Front Med (Lausanne). 2024 Aug 6;11:1430169. doi: 10.3389/fmed.2024.1430169. eCollection 2024. PMID 39165373